CLINICAL TRIAL: NCT05898802
Title: Effect of Kimchi Intake on Body Fat in Overweight Subjects: A Randomized, Double-blind, Placebo-Controlled Trial
Brief Title: Effect of Kimchi Intake on Body Fat in Overweight Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: World Institute of Kimchi (Other Government)
Responsible Party: Principal Investigator, Woo Je Lee, Senior Researcher, World Institute of Kimchi
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: WiKim_2210-037-119
Record Dates: First submitted 2023-06-02; First posted 2023-06-12 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Obesity
Keywords: Kimchi; Lactic acid bacteria
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Participants or study staff working with them will not know what supplements they are receiving.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Kimchi inoculated Leuconostoc mesenteroides (Experimental): 3,600mg/day containing 80% Kimchi inoculated Leuconostoc mesenteroides powder (3 tablets 3 times per day after meals over the 16-week regimen)
  Interventions: Dietary Supplement: Kimchi
- Kimchi (Experimental): 3,600mg/day containing 80% Kimchi powder (3 tablets 3 times per day after meals over the 16-week regimen)
  Interventions: Dietary Supplement: Kimchi
- Lactose (Placebo Comparator): 3,600mg/day containing lactose placebo capsules to look identical. (3 tablets 3 times per day after meals over the 16-week regimen)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Kimchi — Two different kimchi, one traditional kimchi and one fermented with a lactic acid bacteria having anti-obesity effect, hereafter starter kimchi, are flash freeze dried, powdered and encapsulated.
  Arms: Kimchi; Kimchi inoculated Leuconostoc mesenteroides
Dietary Supplement: Placebo — Lactose with kimchi flavor
  Arms: Lactose

SUMMARY:
Kimchi, a traditional Korean food, is prepared through the fermentation of various ingredients. It has been reported that kimchi contains beneficial nutrients from its raw materials, as well as lactic acid bacteria (LAB) and their byproducts produced during fermentation. LAB play an important role in the fermentation process, during which the dominant LAB species emerge and undergo a transition process. Depending on the species and strain of LAB, it has specific functions such as promoting weight loss, reducing inflammation, and lowering cholesterol levels. In this study, the effects of kimchi produced from traditional recipe or kimchi fermented with lactic acid bacteria, which have anti-obesity effects, on body composition changes and metabolic disease index will be investigated in subjects with a BMI of between 23~30kg / m2.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled clinical trial to investigate the anti-obesity effect of kimchi fermented with the addition of specific lactic acid bacteria.

Two different kimchi, one traditional kimchi and one fermented with a lactic acid bacteria having anti-obesity effect, hereafter starter kimchi, are flash freeze dried, powdered and encapsulated. Specifically, subjects with a BMI of between 23~30kg/m2 take 1,200 mg of traditional kimchi or starter kimchi capsules three times per day before each meal, for a total of 3,600 mg per day. As a control, subjects with a BMI of 23 to 30 kg/m2 take lactose capsules in a similar form and in the same amount. The total study period is 16 weeks of intake of kimchi capsules or placebo capsules, excluding the 2 weeks of preparation period for subject selection. Before and after taking the kimchi capsule or the placebo capsule, the following evaluation criteria of the subject will be measured; DEXA (Dual Energy X-ray Absorptiometry), BMI, Weight, Waist to Hip ratio (WHR), total cholesterol, triglyceride, HDL-C, calculate LDL-C, FFA, HbA1c, glucose, insulin, HOMA-IR, hs-CRP, Adiponectin, Leptin. Also, Changes in gut microbiome composition will be determined by measuring bacterial population levels in stool samples collected before and after taking kimchi capsules or placebo capsules.

ELIGIBILITY:
Inclusion Criteria:

* Willing to consent to study participation and to comply with study requirements
* Male and female subjects, 20-65 years of age
* BMI of 23-30 kg/m2
* Those who agreed not to consume Kimchi during the clinical study

Exclusion Criteria:

* Patients with crucial cerebrovascular disease (cerebral infarction, cerebral hemorrhage etc.), or heart failure (angina pectoris, myocardial infarction, heart failure, arrhythmia etc.) or malignancy within 6 months
* Uncontrolled hypertension (Elevated blood pressure (>160/>100))
* Thyroid function test abnormality
* Patients with significantly impaired kidney function: serume creatinine levels ≥2 times upper limit of normal
* Patients with significantly impaired liver function: ALT or AST≥3 times upper limit of normal
* Irregular or occasional gastrointestinal disorders (heartburn, indigestion, etc.)
* Having taken drugs with a known influence on weight in the previous 1 month, such as diet pills, anti-depression drugs, beta-blockers, diuretic, contraceptives, corticosteroids, or female hormones
* Participation in other dietary programmes or services within 3 months
* Participation in other clinical trials within the past 1 month
* Alcohol abuse
* Quitted smoking within 3 months
* Pregnancy or lactation or planning on becoming pregnant
* Have a Kimchi allergy
* Those who are judged unsuitable by the researcher for other reasons
* Taking probiotics within 2 weeks

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2023-07-21 (Actual); Primary Completion 2023-11-09 (Actual); Study Completion 2023-11-09 (Actual)

PRIMARY OUTCOMES:
Fat mass change in 12-week | Baseline (Visit 2, Day 0) and Week 12 (Visit 4, Day 84 ±7)
  Fat mass is measured by DEXA(Dual Energy X-Ray Absorptiometry)

SECONDARY OUTCOMES:
Changes in body mass index (BMI) | Baseline, Week 6, Week 12
  BMI will be calculated as weight (kg) divided by height squared (m²) at baseline, week 6, and week 12.
Changes in body weight | Baseline, Week 6, Week 12
  Body weight will be measured using a calibrated digital scale at baseline, week 6, and week 12.
Changes in waist to hip ratio (WHR) | Baseline, Week 6, Week 12
  Waist to hip ratio will be calculated by dividing waist circumference by hip circumference at baseline, week 6, and week 12.
Changes in Body fat ratio (%) | Baseline and Week 12
  Body fat ratio (%) will be assessed by DEXA
Changes in Body lean mass (kg) | Baseline and Week 12
  Body lean mass (kg) will be assessed by DEXA
Changes in serum lipid profile (Total cholesterol, Triglycerides，Low-density lipoprotein，High density lipoprotein) | Baseline and Week 12
  Fasting blood samples will be collected to measure total cholesterol, triglycerides, LDL-C, and HDL-C at baseline and week 12
Changes in free fatty acids (FFA) concentration | Baseline and Week 12
  Serum free fatty acid concentration will be measured at baseline and week 12.
Changes in HbA1c | Baseline and Week 12
  HbA1c levels will be measured at baseline and week 12 to assess glycemic control.
Changes in fasting glucose concentration | Baseline and Week 12
  Fasting blood glucose concentration will be measured at baseline and week 12.
Changes in insulin resistance | Baseline and Week 12
  Insulin resistance will be assessed using fasting insulin and glucose values at baseline and week 12.
Changes in HOMA-IR value | Baseline and Week 12
  HOMA-IR will be calculated as [fasting insulin (μIU/mL) x fasting glucose (mg/dL)] / 405 at baseline and week 12.
Changes of serum hs-CRP | Baseline and Week 12
  High sensitivity C-reactive protein will be measured at baseline and week 12.
Changes in adiponection | Baseline and Week 12
  Serum adiponectin levels will be measured at baseline and week 12.
Changes in leptin | Baseline and Week 12
  Serum leptin levels will be measured at baseline and week 12.
Change of Microbiota composite | Baseline and Week 12
  Fecal microbiota composition will be assessed at baseline and week 12 using 16S rRNA sequencing.

CONTACTS AND LOCATIONS:
Overall Officials: Wooje Lee, ph.D, Principal Investigator — World Institute of Kimchi; Myungjun Shin, M.D., Ph.D., Study Chair — Pusan National University Hospital
Locations (1):
- Pusan National University Hospital, Busan, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee W, Moon HR, Choi H, Lee HJ, Kim Y, Kim HJ, Yun YR, Kwon MS, Hong SW. Single-cell RNA sequencing reveals that kimchi dietary intervention modulates human antigen-presenting and CD4(+) T cells. NPJ Sci Food. 2025 Nov 17;9(1):236. doi: 10.1038/s41538-025-00593-7. PMID 41249184